CLINICAL TRIAL: NCT02585362
Title: Influence of a Specially Formulated Whey Protein Supplement in Combination With Physical Exercise and Nutrition Program on Physical Performance in Cancer Outpatients
Brief Title: Whey Protein Supplement in Combination With Physical Exercise and Nutrition Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kantonsspital Winterthur KSW (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Leucine1.0
Record Dates: First submitted 2015-10-13; First posted 2015-10-23 (Estimated); Last update posted 2019-01-11 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer; Gastro-Intestinal Cancer; Breast Cancer; Prostate Cancer; Pleural Mesothelioma; Urothelial Carcinoma; Renal Cell Carcinoma; Ovarian Cancer
Keywords: palliative
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Prostatic Neoplasms; Mesothelioma, Malignant; Carcinoma, Transitional Cell; Carcinoma, Renal Cell; Ovarian Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Active Comparator): Participants will receive physical exercise, nutrition counseling and a whey protein Supplement over 12 weeks
  Interventions: Behavioral: physical exercise; Behavioral: nutrition counseling; Dietary Supplement: whey protein supplement
- Control group (No Intervention): Participants will receive standard care

INTERVENTIONS:
Behavioral: physical exercise — The standardized Training program will be performed twice a week in the Kantonsspital Winterthur and once a week in a home based setting
  Arms: Intervention group
Behavioral: nutrition counseling — At least 3 times, participants will receive nutrition counseling to improve energy- and protein intake
  Arms: Intervention group
Dietary Supplement: whey protein supplement — On workout days study participants will consume twice a day 15 g of the supplement powder with approximately 150 ml water. On the remaining days participants consume the supplement once a day.
  Arms: Intervention group

SUMMARY:
This study evaluates physical performance in cancer outpatients during a multimodal therapy. Half of the patients will receive physical exercise und nutrition program in combination with a specially formulated whey protein supplement, while the other half will receive standard care.

DETAILED DESCRIPTION:
The time period of Intervention will last 3 month, measurements will be conducted at baseline and 3 month. After 6 month there will be an additional follow-up test point to assess the sustainability of the intervention. The 3-month intervention study consists of a physical exercise program and nutrition counseling in combination with a specially formulated whey protein supplement high in leucine. The standardized training program will be performed twice a week in the physical department of the Kantonsspital Winterthur (KSW) and once a week in a home based setting. Additionally, participants of the intervention group will be aks to consume 15 g of the nutrient supplement powder with approximately 150 ml water. On workout days the supplement should be taken twice a day and on the remaining days once a day. During the three month intervention study participants will take part in a nutrition counseling for at least three times.

ELIGIBILITY:
Inclusion Criteria:

* Advanced cancer patients not eligible for curative treatment: lung cancer, gastrointestinal cancer, breast cancer, prostate cancer, ovarian cancer, pleural mesothelioma, urothelium carcinoma, renal cell carcinoma
* WHO performance status ≥ 2
* Able to walk independently at least 100 meters
* Estimated life expectancy of ≥ 6 month

Exclusion Criteria:

* Patients currently using nutritional supplements with branched chain amino acids
* Enteral or parenteral nutrition within 1 month
* History of ileus within 1 month
* Psychiatric disorder precluding understanding of information on trials related topics and giving informed consent
* Milk protein allergy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

PRIMARY OUTCOMES:
Change in physical performance | measured at week 0, 12 and 24
  Physical performance will be assessed with the short physical performance battery

SECONDARY OUTCOMES:
Change in body composition | measured at week 0, 12 and 24
  Body composition will be assessed with bioimpedance
Change in quality of life | measured at week 0, 12 and 24
  Quality of life will be assessed with the questerionnaire EORTC-QLQ-C30
Change in fatigue | measured at week 0, 12 and 24
  Fatigue will be assessed with the questionnaire brief fatigue inventory
Change in physical function | measured at week 0, 12 and 24
  Physical function will be assessed with 60s-sit-to-stand-test and timed-up&go-test
Change in nutritional status | measured at week 0, 12 and 24
  Nutritional status will be assessed with hand grip, nutritional risk screening 2002 and patient-generated subjective global assessment
Change in diet history | measured at week 0, 12 and 24
  3-day food records brought in at weeks 0, 12 and 24 will be analyzed for energy- and protein intakes
Number of re-hospitalization | up to 24 weeks
  Number of re-hospitalization
Change in WHO performance status | measured at week 0, 12 and 24
  Change in WHO performance status
Overall survival | up to 24 weeks
  Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Miklos Pless, Prof., Principal Investigator — Kantonsspital Winterthur KSW
Locations (1):
- Kantonsspital Winterthur, Winterthur, Switzerland

IPD SHARING:
Plan to Share IPD: No